CLINICAL TRIAL: NCT05625542
Title: RELIEF CENSUS-US: Cross-sectional Study to Assess Prevalence and Burden of CKD-associated Pruritus in Hemodialysis Patients
Brief Title: Cross-sectional Study to Assess Prevalence and Burden of CKD-associated Pruritus in Hemodialysis Patients
Acronym: CKD
Status: Withdrawn | Type: Observational
Why Stopped: The study will not be conducted
Sponsor: Vifor (International) Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Other Study IDs: CS-DFK-2022-0027
Record Dates: First submitted 2022-11-01; First posted 2022-11-23 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Chronic Kidney Disease-associated Pruritus
Keywords: CKD; CKD-AP; CKD associated pruritus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Vifor International Ltd. is seeking real-world evidence (RWE) to better understand the epidemiology, patient characteristics, and management of CKD-aP in the real-world clinical setting.

DETAILED DESCRIPTION:
CKD-aP is a global clinical problem, and finding effective treatment remains a therapeutic challenge because of its complex pathophysiology (Sommer 2007, Weisshaar 2019, Yosipovitch 2013). The association between CKD-aP and clinical features and laboratory data remains unclear (Davison 2021, Manenti 2021). CKD-aP is thought to be associated with several conditions, including vitamin D deficiency, metabolic abnormalities (e.g., abnormal serum calcium or phosphate levels), toxin build-up, peripheral neuropathy, immune system dysregulation, or opioid receptor dysregulation (Jung 2015, Xie 2021, Kremer 2019, Verduzco 2020, Swarna 2019, Manenti 2021).

At present, there is no systematic assessment of CKD-aP in routine clinical practice, and the prevalence of CKD-aP is generally under-reported by patients and therefore underestimated by as much as 69% of healthcare professionals (HCPs) (Rayner 2017). Alleviating the burden of CKD-aP requires proactive identification of patients who suffer from it (Sukul 2020, Davison 2015, Phan 2012).

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patients with CKD (≥18 years) receiving HD for at least 3 months prior to signing informed consent
* Signed informed consent
* Able and willing to fill in questionnaires

Exclusion Criteria:

* Patients receiving HD at home or both home and site

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — male or female adult patients (≥18 years) undergoing HD
Study Population: The study will consist of a random selection of approximately 3,330 male or female adult patients (≥18 years) undergoing HD within two large dialysis organization (DO) networks.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence (%) of CKD-aP patients undergoing HD based on the WI-NRS score (past 24 hours). | Day 1
  Ratio between the overall number of patients with WI-NRS scores ranging from 1-10 and the overall number of patients with WI-NRS scores ranging from 0-10, from patients randomly selected to participate in the study.

SECONDARY OUTCOMES:
Prevalence (%) of patients undergoing HD with various CKD-aP severities based on the WI-NRS score (past 24 hours). | Day 1
  none (0), mild (1-3), moderate (4-6), or severe (7-10) scores
Current socio-demographic, clinical, and dialysis characteristics as well as current therapeutic landscape | Day 1
  in the management of CKD-aP
Impact of pruritus severity (WI-NRS)on HRQoL, | Day 1
  as reported by patients
Patient-reported communication with physician and other healthcare provider with respect to pruritus, as well as self-reported anti-itch treatments. | Day 1
  Pruritus and anti-itch
Clinical and healthcare resource outcomes in the last 12 months. | Day 1
  Missed or additional dialysis sessions, Hospitalizations, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Despina Rüssmann, Dr, Study Chair — CSL Vifor

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement
Supporting Information: Study Protocol, SAP
Time Frame: Data can be requested 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later.
Access Criteria: A research proposal must be approved by an independent review panel and the study sponsor and researchers must sign a data sharing agreement.